CLINICAL TRIAL: NCT00203619
Title: An Economic Evaluation of Capsule Endoscopy for Obscure Gastrointestinal Bleeding
Brief Title: Capsule Endoscopy in Obscure GI Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Heritage Foundation for Medical Research (Other); Calgary Health Region (Other)
Responsible Party: Principal Investigator, Dr. Robert Hilsden, Associate Professor, Department of Medicine & Research Director, Colon Cancer Screening Centre, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Obscure Gastrointestinal Bleeding
MeSH Terms: interventions — Capsule Endoscopy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Wireless capsule endoscopy
  Interventions: Device: Wireless capsule endoscopy
- 2 (Active Comparator): Standard care
  Interventions: Other: standard care

INTERVENTIONS:
Device: Wireless capsule endoscopy — wire less capsule endoscopy
  Arms: 1
Other: standard care — standard diagnostic evaluation as decided by treating physician
  Arms: 2

SUMMARY:
The purpose of this study is to conduct a cost-effectiveness analysis of wireless capsule endoscopy in the investigation of patients with overt obscure gastrointestinal bleeding. To inform this analysis, a randomized controlled trial of capsule endoscopy compared with standard care will be conducted

DETAILED DESCRIPTION:
The purpose of this study is to conduct a cost-effectiveness analysis of wireless capsule endoscopy in the investigation of patients with overt obscure gastrointestinal bleeding. To inform this analysis, a randomized controlled trial of capsule endoscopy compared with standard care will be conducted. Patients randomized 1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Obscure overt GI bleeding
3. No cause for bleeding found on Gastroscopy and colonoscopy within 1 week of bleeding

Exclusion Criteria:

1. Known or suspected swallowing disorders
2. Known or suspected small bowel obstruction
3. Multiple comorbidities precluding surgery
4. Patients with implantable electromagnetic devices
5. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-05; Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
sf36 | 48 weeks
giqli | 48 weeks
eq50 | 48 weeks
diagnostic yield | 48 weeks

SECONDARY OUTCOMES:
transfusions | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Hilsden, MD PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada